CLINICAL TRIAL: NCT05595291
Title: Walking Characteristics of Patients With Amputation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associate Professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 29
Record Dates: First submitted 2022-10-22; First posted 2022-10-26 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Amputation
Keywords: amputation; walking; satisfaction; pain
MeSH Terms: conditions — Personal Satisfaction; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: investigation of the factors affecting walking characteristics — In order to investigate the factors affecting walking characteristics, 2-minute walking test, 10-point VAS (overall prosthesis satisfaction level, socket comfort and satisfaction level, knee joint satisfaction level, prosthetic foot satisfaction level, pain level in amputated extremity) and locomotor capacity index will be applied.

SUMMARY:
The main purpose of the study is to reveal the early and late changes in the walking characteristics of patients with lower extremity amputation. Secondly, it is planned to reveal the factors affecting the walking characteristics of patients with amputation and to compare individuals with different levels of amputation in terms of clinical outcome measures.

DETAILED DESCRIPTION:
It is important to investigate the long-term changes in walking characteristics of patients with amputation and the factors affecting walking characteristics in these patients regarding prosthesis rehabilitation.

The main purpose of the study is to reveal the early and late changes in the walking characteristics of patients with lower extremity amputation. Secondly, it is planned to reveal the factors affecting the walking characteristics of patients with amputation and to compare individuals with different levels of amputation in terms of clinical outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65
* Presence of lower extremity amputation

Exclusion Criteria:

* Conditions that prevent the use of prosthesis (wound, pain, etc.)
* Having a history of rheumatic disease
* Having cardiac pathology
* Having pulmonary pathology
* Having a situation that prevents communication
* Not giving written consent

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred patients with lower extremity amputation will be participated in this cross-sectional study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-05 (Estimated); Primary Completion 2023-02-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
2-minute walking test | through study completion, an average of one month
  Walking distance will be evaluated using the two-minute walking test (2MWT). Patients will be instructed to walk quickly, safely, and as much distance as possible along a rectangular path.

SECONDARY OUTCOMES:
Visual Analog Scale | through study completion, an average of one month
  All patients will mark the severity of amputated extremity pain on a Visual Analog Scale (VAS; from 0 (no pain) to 10 (worst pain)). The socket system comfort and satisfaction, knee joint satisfaction, prosthetic foot satisfaction and overall prosthesis satisfaction will be evaluated with a 10-point VAS (from 0 (absolutely dissatisfied) to 10 (absolutely satisfied)).
Locomotor capacity index | through study completion, an average of one month
  The Locomotor Capabilities Index (LCI) is a validated measure of lower-limb amputees' ability to perform activities with prosthesis. The total LCI score is the sum of the item scores and can range from 0 (worst) to 30 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Demir, Principal Investigator — Associate Professor